CLINICAL TRIAL: NCT03261115
Title: Efficacy of Topical Benzocaine in Anterior Maxilla: A Randomised Controlled Trial
Brief Title: Effects of Benzocaine 20% Topical Anesthetic and no Topical Agent on Pain Perception During Intra-oral Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nurain Rehman (Other)
Responsible Party: Sponsor-Investigator, Nurain Rehman, Final Year Student BDS, CMH Lahore Medical College and Institute of Dentistry
Organization: CMH Lahore Medical College and Institute of Dentistry (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NR3517
Record Dates: First submitted 2017-08-18; First posted 2017-08-24 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Anesthesia
Keywords: Pain, Benzocaine, Clinical trial
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Topical Anesthesia
- Study group (Experimental): No topical anesthesia
  Interventions: Procedure: No topical anesthesia

INTERVENTIONS:
Procedure: No topical anesthesia — Lack of use of topical anesthesia application prior to infiltration injection intra-orally
  Arms: Study group

SUMMARY:
The aim of this randomized controlled trial. is to test the efficacy of topical anesthesia against the use of no topical agent during buccal infiltration in maxillary anterior teeth. The rationale behind this comparison is to evaluate the practical, clinical outcome of not using any topical agent if in fact topical anesthesia does not reduce pain as reported by various studies and if consequently its usage was to be discontinued.

DETAILED DESCRIPTION:
The clinical implication of topical anesthesia and placebo being the same is to not use either of them prior to LA administration in dentistry. This clinical approach has rarely been studied and this study aims to compare the effects of the use of topical anesthesia against the use of no topical agent prior to buccal infiltration in maxillary anterior teeth.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18
* Males and females both
* Participants requiring extraction of maxillary anterior teeth
* Intact or minimally restored anterior teeth
* Patients with American Society of Anesthesiologists physical status of 1 or 2

Exclusion Criteria:

* Participants with physical American Society of Anesthesiologists physical status of 3 or 4
* Showing signs of inflammation in the area to be injected
* Having known allergy to any of the agents used in the study
* Used anti- anxiety drugs or sedatives in the past two weeks
* Have taken analgesics on the day of data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2017-09-16 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Pain score on needle penetration | Immediately
  Pain score measured by numeric pain rating scale
Pain score on local anesthesia deposition | Immediately
  Pain score measured by numeric pain rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Nurain Rehman, Principal Investigator — CMH Lahore Medical College and Institute of Dentistry; Samir Qazi, FFDRCSI, Study Director — CMH Lahore Medical College and Institute of Dentistry
Locations (1):
- CMH Lahore Medical College and Institute of Dentistry, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rehman N, Qazi SR. Efficacy of Topical Benzocaine in Maxilla: A Randomized Controlled Trial. Anesth Prog. 2019 Spring;66(1):24-29. doi: 10.2344/anpr-66-01-01. PMID 30883233